CLINICAL TRIAL: NCT05813236
Title: Randomized, Monocentric, Double Blinded, Prospective Study to Evaluate the Early Wound Healing After the Utilization of NOVOSYN® Quick Versus MONOSYN® Quick Suture Material in Resective Periodontal Surgery
Brief Title: NOVOSYN® Quick Versus MONOSYN® Quick Suture Material in Resective Periodontal Surgery
Acronym: NOQMOQS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAG-O-H-2109
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Gingivitis; Gingival Diseases; Periodontal Diseases
Keywords: Resective periodontal surgery
MeSH Terms: conditions — Gingivitis; Gingival Diseases; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Patients undergoing resective periodontal surgery will randomly (1:1) receive Novosyn Quick (control group) or Monosyn Quick (treatment group).
  Randomization will take place intraoperatively through dynamic allocation with minimisation algorithm to a suture group. Randomization will be stratified by study site.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and the observers (assessors) will be blinded to the applied suture material.
  Patients will not be informed which suture material will be applied. The observers (assessors) who will perform the assessment of the wounds will also be unaware of the applied suture type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novosyn® (Experimental): Novosyn® Quick is available in a range of gauge sizes and lengths, non-needled or attached to stainless steel needles of varying types and sizes: Novosyn® Quick sutures are available undyed in sizes USP 2 (5 metric) through USP 6-0 (0.7 metric).
  Interventions: Device: Novosyn® in resective periodontal surgery
- Monosyn® (Active Comparator): Monosyn® Quick is a sterile, synthetic, absorbable, monofilament surgical suture material made from a triblock copolymer comprising glycolide (72 %), ε-caprolactone (14 %) and trimethylene carbonate (14 %), which is only available undyed.
  Interventions: Device: Monosyn® in resective periodontal surgery

INTERVENTIONS:
Device: Novosyn® in resective periodontal surgery — The aim of resective procedures is the re-establishment of a healthy periodontium at a reduced level, accepting as irreversible the destruction that has already occurred. In essence, these procedures are all designed to achieve pocket elimination or reduction by the apical shift of the gingival margin.
  Arms: Novosyn®
Device: Monosyn® in resective periodontal surgery — The aim of resective procedures is the re-establishment of a healthy periodontium at a reduced level, accepting as irreversible the destruction that has already occurred. In essence, these procedures are all designed to achieve pocket elimination or reduction by the apical shift of the gingival margin.
  Arms: Monosyn®

SUMMARY:
The aim of this study is to prove that Novosyn Quick and Monosyn Quick are equivalent in early wound healing in adult patients undergoing resective periodontal surgery.

In order to show equivalence between Novosyn Quick and Monosyn Quick EHS, which is composed of 3 parameters: clinical signs of reepithelization, clinical signs of haemostasis and clinical signs of inflammation, will be calculated for each suture 10 ± 5 days postoperatively and cannot differ more than 2 points.

Furthermore, complications, the handling of the suture material, pain, satisfaction of the patient and bacterial contamination of the thread (optional) will also be assessed as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing resective periodontal surgery abd one of the incisions below has been performed:
* Crestal incision
* Vertical incision
* Intrasulcular incision
* Submarginal incision
* Written informed consent regarding the data collection for the RCT

Exclusion Criteria:

* Emergency surgery.
* Pregnancy.
* Breastfeeding
* Patients taking medication that might affect wound healing.
* Patients having a condition that might affect wound healing.
* Patients with hypersensitivity or allergy to the suture material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
early wound healing score (EHS) | 10 ± 5 days postoperatively
  The primary end point in order to evaluate the primary objective of the study will be the determination of early wound healing score (EHS) in patients undergoing resective periodontal surgery. The EHS will be evaluated in 3 parameters: clinical signs of re-epithelization (CSR), clinical signs of haemostasis (CSH), and clinical signs of inflammation (CSI). Zero, 3 or 6 points have been used to evaluate the CSR, whereas 0, 1, or 2 points have been used for both CSH and CSI (Table 3). The summation of these 3 parameters generated the EHS. The EHS for ideal wound healing was 10 points, while the worst possible score was 0 points. An EHS of 0 points was assigned in the presence of suppuration, independently of the ratings for the 3 single parameters.

SECONDARY OUTCOMES:
Number of patients showing postoperative wound dehiscence | 10 ± 5 days postoperatively
  Incidence of wound dehiscence after resective periodontal surgery. Dehiscence is the
Number of patients showing postoperative Dentinal hypersensitivity | 10 ± 5 days postoperatively
  Incidence of Dentinal hypersensitivity after resective periodontal surgery
Number of patients showing postoperative Oral candidiasis | 10 ± 5 days postoperatively
  Incidence of oral candidiasis after resective periodontal surgery
Number of patients showing postoperative Angular cheilitis | 10 ± 5 days postoperatively
  Incidence of Angular cheilitis after resective periodontal surgery
Number of patients showing postoperative Swelling | 10 ± 5 days postoperatively
  Incidence of Swelling after resective periodontal surgery
Number of patients showing postoperative Bleeding | 10 ± 5 days postoperatively
  Incidence of Bleeding after resective periodontal surgery
Number of patients showing postoperative Infection | 10 ± 5 days postoperatively
  Incidence of infection after resective periodontal surgery
Number of Systemic complications | 10 ± 5 days postoperatively
  The number of systemic complications is summarized, this includes fever, skin rash, neuropraxia, trismus, osteomyelitis, sinusitis and other complications.
Pain assessment | 10 ± 5 days postoperatively
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal pain"
Satisfaction of the patient | 10 ± 5 days postoperatively
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "not satisfied at all" and "100" at the opposite end representing "completely satisfied"
Number of patients with Bacterial contamination of the thread (optional) | 10 ± 5 days postoperatively
  Assessment of bacterial colonization on the thread of the suture will be evaluated by sending the swab of the suture to laboratory to be investigated and analysed. Polymerase Chain Reaktion Test (PCR) analysis is the test used for bacterial colonization. The micro-IDent® and micro-IDent® plus tests are able to identify 11 bacterial pathogens, including two complex pathogens.
Assessment of the handling of the suture material | intraoperatively
  Assessment of the suture material will be performed intra-operatively using a questionnaire including different dimensions (ease of passage through the tissue, first throw knot holding, knot security, knot tie down smoothness, surgical hand, memory effect and degree of fraying) with 5 point scale (excellent, very good, good, satisfied, poor) and the overall handling of the suture material.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Mor Reinoso, Dra., Principal Investigator — Facultat d'Odontologia. Universitat Internacional de Catalunya
Locations (1):
- Facultat d'Odontologia. Universitat Internacional de Catalunya, Sant Cugat del Vallès, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No